CLINICAL TRIAL: NCT00133211
Title: Medical Antiarrhythmic Treatment or Radiofrequency Ablation in Paroxysmal Atrial Fibrillation: A Randomized Prospective Multicentre Study (MANTRA-PAF)
Brief Title: Radiofrequency Ablation (RFA) Versus Antiarrhythmic Drug Treatment in Paroxysmal Atrial Fibrillation
Acronym: MANTRA-PAF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Danish Heart Foundation (Other)
Responsible Party: Principal Investigator, Jens Cosedis Nielsen, MD, DMSc, associate professor, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sks2005psh01; NCT00133211
Record Dates: First submitted 2005-08-22; First posted 2005-08-23 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Atrial Fibrillation
Keywords: Paroxysmal atrial fibrillation; Heart arrhythmia; Ablation; Drug treatment
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Antiarrythmic drug treatment
  Interventions: Procedure: Radiofrequency ablation
- 2 (Experimental)
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Radiofrequency ablation — Pulmonary vein isolation

SUMMARY:
Atrial fibrillation is the most common heart arrhythmia afflicting approximately 1% of the Danish population. Medical antiarrhythmic treatment is only moderately effective and has the risk of severe side effects. The present study is a prospective, randomized, multicentre study comparing medical antiarrhythmic drug strategy with catheter based radiofrequency strategy in patients with paroxysmal atrial fibrillation. The primary end point is atrial fibrillation burden (symptomatic and asymptomatic) judged by multiple 7-day Holter monitorings during 2 years follow-up. Three hundred patients considered candidates for antiarrhythmic drug treatment will be randomized. The study will be performed as a Scandinavian/German multicentre study.

DETAILED DESCRIPTION:
Introduction:

Atrial fibrillation is by far the most common heart arrhythmia and is even increasing in prevalence and incidence. Approximately 10% of all cardiologic hospitalizations are due to atrial fibrillation. Several studies have shown older patients with paroxysmal or persistent atrial fibrillation and with minor symptoms related to the arrhythmia do equally well on a frequency control as compared to a rhythm control strategy. However, some of this lack of difference in outcome may be because the benefits by achieving sinus rhythm are outbalanced by the risk of medication with presently known antiarrhythmic drugs together with the only modest efficacy of these drugs. Non-pharmacological treatment of atrial fibrillation has drawn increasing interest over the last decade, and especially percutaneous catheter based ablation strategies have been in focus with promising results on the symptomatic level in several series of patients. Different technologies have been in use with very few comparative studies. Most important, no study has been published so far on a consecutive series of patients with atrial fibrillation randomized to either a pharmacological or an ablative strategy. Also important is that the majority of studies have been single-centre based prone to a multitude of potential selection biases.

Hypothesis:

Pulmonary vein isolation by transvenous radiofrequency ablation is superior to present time antiarrhythmic drug therapy with regard to long-term suppression of atrial fibrillation (symptomatic and asymptomatic) as well as to procedure/treatment related side effects.

Purpose:

The present study is designed to test whether catheter based radiofrequency ablation is superior to optimized antiarrhythmic medical therapy in suppressing long-term relapse of symptomatic and/or asymptomatic atrial fibrillation in patients who are not already in chronic pharmaceutical antiarrhythmic therapy. Secondary end points are: mortality, thromboembolic events, hospitalization due to disturbance in heart rhythm, proarrhythmic events, procedure/treatment related side effects, health economics and quality of life. Comparison will be made after two years follow-up and a register follow-up will take place after additional 3 years (a total of at least five years of follow-up).

Consecutive patients fulfilling the inclusion criteria will be informed about the study by a study-responsible electrophysiologist or his/her substitute. After informed consent the patient will be randomized to either antiarrhythmic drug treatment or to catheter ablation. All patients undergo transthoracic echocardiography before randomization.

A register of all patients informed about (i.e. fulfilling the inclusion criteria) but for one or more reasons not included in the study will be established.

Primary endpoint:

Atrial fibrillation burden (see below), symptomatic and asymptomatic combined. Atrial fibrillation burden will be calculated from one-week Holter monitoring at 3, 6, 12, 18 and 24 months, respectively, after treatment (first RF-procedure or AAD-initiation).

Secondary endpoints:

* Mortality
* Complications (including thromboembolic events, major bleeding episodes, pro-arrhythmic events, and treatment related side effects)
* QOL
* Health economics (including number of DC-conversions, cardiovascular hospitalizations (type, length and number of antiarrhythmic drugs))
* Chronic atrial fibrillation (constant atrial fibrillation during one-week Holter monitoring at 24 months follow-up, together with atrial fibrillation during the immediately foregoing 8 weeks)
* Time to first recurrence (after 3 months blanking period)
* Left ventricular systolic function (transthoracic echo)

ELIGIBILITY:
Inclusion Criteria:

* Patients ≤ 70 years of age
* Paroxysmal atrial fibrillation patients who are considered as being candidates for antiarrhythmic drug therapy initiation
* Patients who have had at least two episodes of symptomatic paroxysmal atrial fibrillation in the foregoing 6 months can be included. The atrial fibrillation episodes may be persistent (need DC- or AAD-conversion) with a duration of less than 7 days.

Exclusion Criteria:

* Previous or ongoing chronic treatment with class IC or class III antiarrhythmic drugs
* Intolerance/contraindication to class IC and class III antiarrhythmic drugs (i.e. intolerance/contraindication to only one of the two groups is not excluding the patient)
* Previous atrial fibrillation ablation
* Severely increased left atrial size
* Left ventricular ejection fraction below 0.40 (during sinus rhythm or atrial fibrillation with RR-intervals above 600 ms) or "eye-balled" reduction of systolic function to less than "moderately decreased".
* Contraindication to anticoagulation treatment with vitamin K antagonists
* Expected surgery for structural heart disease within the follow-up period Significant mitral valve disease
* New York Heart Association (NYHA) III-IV
* Planned pregnancy within the follow-up period
* Secondary atrial fibrillation (e.g. post-surgery, infections, hyperthyroidism)
* Age < 18 years
* Patient does not want to participate.

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2005-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation burden | Two years

SECONDARY OUTCOMES:
mortality | 2 years
complications to treatment | 2 years
Quality of life | 2 years
Health economics | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jens Cosedis Nielsen, MD, DMSc, Principal Investigator — Aarhus University Hospital Skejby
Locations (1):
- Department of Cardiology, Aarhus, Denmark

REFERENCES:
- [Derived] Nielsen JC, Johannessen A, Raatikainen P, Hindricks G, Walfridsson H, Pehrson SM, Englund A, Hartikainen J, Mortensen LS, Hansen PS; MANTRA-PAF Investigators. Long-term efficacy of catheter ablation as first-line therapy for paroxysmal atrial fibrillation: 5-year outcome in a randomised clinical trial. Heart. 2017 Mar;103(5):368-376. doi: 10.1136/heartjnl-2016-309781. Epub 2016 Aug 26. PMID 27566295
- [Derived] Walfridsson H, Walfridsson U, Nielsen JC, Johannessen A, Raatikainen P, Janzon M, Levin LA, Aronsson M, Hindricks G, Kongstad O, Pehrson S, Englund A, Hartikainen J, Mortensen LS, Hansen PS. Radiofrequency ablation as initial therapy in paroxysmal atrial fibrillation: results on health-related quality of life and symptom burden. The MANTRA-PAF trial. Europace. 2015 Feb;17(2):215-21. doi: 10.1093/europace/euu342. Epub 2015 Jan 6. PMID 25567068
- [Derived] Aronsson M, Walfridsson H, Janzon M, Walfridsson U, Nielsen JC, Hansen PS, Johannessen A, Raatikainen P, Hindricks G, Kongstad O, Pehrson S, Englund A, Hartikainen J, Mortensen LS, Levin LA. The cost-effectiveness of radiofrequency catheter ablation as first-line treatment for paroxysmal atrial fibrillation: results from a MANTRA-PAF substudy. Europace. 2015 Jan;17(1):48-55. doi: 10.1093/europace/euu188. Epub 2014 Oct 23. PMID 25341739
- [Derived] Cosedis Nielsen J, Johannessen A, Raatikainen P, Hindricks G, Walfridsson H, Kongstad O, Pehrson S, Englund A, Hartikainen J, Mortensen LS, Hansen PS. Radiofrequency ablation as initial therapy in paroxysmal atrial fibrillation. N Engl J Med. 2012 Oct 25;367(17):1587-95. doi: 10.1056/NEJMoa1113566. PMID 23094720